CLINICAL TRIAL: NCT05008549
Title: A Randomized, Double-blinded, Placebo-controlled, Crossover Study, to Assess the Synergistic Effects of a Cranberry Beverage on Cognitive Function
Brief Title: A Study to Assess the Synergistic Effects of a Cranberry Beverage on Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ocean Spray Cranberries, Inc. (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: AFCRO-140
Record Dates: First submitted 2021-07-14; First posted 2021-08-17 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Attention; Mood
MeSH Terms: interventions — theanine

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded, placebo-controlled, crossover study, to assess the synergistic effects of a cranberry beverage on cognitive function in healthy adults aged 18-45.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- First Product Order: order not stated to protect study blinding (Experimental): Participants will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for 7 days, followed by a 7 day wash-out period before beginning the next product in the sequence.
  Interventions: Dietary Supplement: Cranberry Juice Product
- Second Product Order: order not stated to protect study blinding (Experimental): Participants will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for 7 days, followed by a 7 day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Cranberry Juice Product
- Third Product Order: order not stated to protect study blinding (Experimental): Participants will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for 7 days, followed by a 7 day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Cranberry Juice Product
- Fourth Product Order: order not stated to protect study blinding (Experimental): Participants will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for 7 days, followed by a 7 day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Cranberry Juice Product
- Fifth Product Order: order not stated to protect study blinding (Experimental): Participants will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for 7 days, followed by a 7 day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Cranberry Juice Product
- Sixth Product Order: order not stated to protect study blinding (Experimental): Participants will receive each of the 6 study products sequentially in a cross-over design, consuming one study product for 7 days, followed by a 7 day wash-out period before beginning the next product in the sequence
  Interventions: Dietary Supplement: Cranberry Juice Product

INTERVENTIONS:
Dietary Supplement: Cranberry Juice Product — The cranberry juice product contains 100 % cranberry juice (ingredients: water, cranberry juice concentrate)
  The cranberry juice + lemon balm extract product contains 100 % cranberry juice (ingredients: water, cranberry juice concentrate) + lemon balm extract (300 mg, Robertet Groupe)
  The cranberry juice + tart cherry juice product contains 100 % cranberry juice (ingredients: water, cranberry juice concentrate) + 3 g tart cherry powder (Cherry PURE)
  The cranberry juice + L-theanine product contains 100% cranberry juice (ingredients: water, cranberry juice concentrate) + 200 mg L-theanine (Suntheanine, Taiyo International)
  L-theanine + placebo product contains L-theanine (200 mg, Suntheanine, Taiyo International) + placebo (see 5.2.1)
  The placebo product contains water, dextrose, citric acid, malic acid, fumaric acid, natural flavor, Red #40, xanthan gum, Blue #1, gum Arabic, Reb M, Steviol glycosides, and ester gum.
  Other Names: Cranberry Juice + Lemon Balm Extract Product; Cranberry Juice + Tart Cherry Juice Product; Cranberry Juice + L-theanine Product; L-theanine + Placebo Product; Placebo Product

SUMMARY:
This study aims to determine the effect short-term dosing (7 days) of a placebo beverage, cranberry juice, cranberry juice + lemon balm extract, cranberry juice + tart cherry powder, or cranberry juice + L-theanine or L-theanine beverage on cognitive function and mood in healthy adults (18-45 years). The study will include measures of attention, alertness, performance, and mood/stress.

DETAILED DESCRIPTION:
1.1 Background information Berries from the Vaccinium genus have been reported to improve some measures of cognitive function in healthy adults. There is evidence that the polyphenols contained in berries and other plant foods may play a role in this regard. Among the plant sources of polyphenols, lemon balm and tart cherry reported to have positive effects on cognitive function in randomized controlled trials (RCTs).

L-theanine is an amino acid present almost exclusively in the tea plant (Camellia sinesis). L-theanine crosses the blood-brain barrier and has been shown to increase serotonin and dopamine production in rats. A recent systematic review of RCTs that evaluated the effect of supplemental L-theanine on stress concluded that L-theanine may assist in the reduction of stress.

Given that plant bioactives may have varying mechanisms to support cognitive health, the aim of this study is as follows:

Aim 1: To determine the effect short-term dosing (7 days) of a placebo beverage, cranberry juice, cranberry juice + lemon balm extract, cranberry juice + tart cherry powder, or cranberry juice + L-theanine or L-theanine beverage on cognitive function and mood in healthy adults (18-45 years). The study will include measures of attention, alertness, performance, and mood/stress.

1.2 Investigational product

Beverage to be tested:

* 100% cranberry juice (8 oz, Ocean Spray)
* 100% cranberry juice (8 oz) + lemon balm extract (300 mg)
* 100% cranberry juice (8 oz) + tart cherry powder (3 g)
* 100% cranberry juice (8 oz) + L-theanine (200 mg)
* L-theanine (200 mg) + placebo (matched for color, taste, calories)
* placebo (matched for color, taste, calories) 1.3 Rationale for conducting the clinical trial There is scientific support for Vaccinium berries to be of benefit to cognitive health. However, this has not be specifically tested in cranberries (Vaccinium macrocarpon). Furthermore, the individual effects of the other ingredients to be tested in this trial have been found to have positive effects on cognitive health but whether there are added effects with cranberry is not known.

  2 OBJECTIVES 2.1 Primary objective To evaluate in healthy adults the effect of 7-day consumption of cranberry beverages compared to placebo on attention.

2.2 Primary endpoint variable

* Change in Accuracy of Attention composite scores outcomes from Baseline to each treatment phase (V3-8), assessed using the COMPASS cognitive assessment tool.
* Change in Speed of Attention composite scores outcomes from Baseline to each treatment phase (V3-8), assessed using the COMPASS cognitive assessment tool.

2.3 Secondary objectives To evaluate in healthy adults the effect of 7-day consumption of cranberry beverages compared to placebo on measures of focus, alertness, and cognition.

To evaluate in healthy adults the effect of 7-day consumption of cranberry beverages compared to placebo on mood and stress.

2.4 Secondary endpoint variables

* Focus: Change in Overall % accuracy scores outcomes from Baseline to each treatment phase (V3-8), assessed using the STROOP task in the COMPASS cognitive assessment tool.
* Alertness: Change in Alertness scores outcomes from Baseline to each treatment phase (V3-8), assessed using the self-rated Alertness VAS scale in the COMPASS cognitive assessment tool.
* Cognitive Performance:

  * Change in Accuracy of Performance composite scores outcomes from Baseline to each treatment phase (V3-8), assessed using the COMPASS cognitive assessment tool.
  * Change in Speed of Performance composite scores outcomes from Baseline to each treatment phase (V3-8), assessed using the COMPASS cognitive assessment tool.
* Mood: Change in Total Mood Disturbance scores from Baseline to each subsequent visit (V3-8), assessed using the Profile of Mood States-Short Questionnaire.
* Stress: Change in salivary cortisol from Baseline to each treatment phase (V3-8).

2.5 Exploratory objectives Dependent upon the outcome of the Primary and Secondary objectives, additional outcomes from the COMPASS cognitive assessment tool may be analyzed further to assess the impact of the investigational product on various domains of cognition.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion, the participant must fulfil all of the following criteria:

1. Be able to give written informed consent and willing/able to comply with study procedures.
2. Be between 18 and 45 years, inclusive.
3. Is in general good health, as determined by the investigator.
4. Has a BMI between ≥20 - ≤35 kg/m2.
5. Has had a stable body weight (≤5 % change) over the past 3-months.
6. Has a Beck Depression Inventory II score ≤20 at screening.
7. Willing to discontinue consumption of wine and dark red/blue colored fruits and polyphenol-rich fruits (e.g., pomegranate, blueberries, grapes), lemon balm, tart cherry powder, and L-Theanine for the two weeks leading up to the study (from the Screening visit V1 to baseline V2) and during the study.
8. Willing and able to avoid consumption of any cranberry juice, whole cranberries, and dried cranberries for the two weeks leading up to the study (from the Screening visit V1 to baseline V2) and during the study, excluding the study beverage.
9. Is willing to provide saliva samples.
10. Maintain current level of physical activity and dietary habits throughout the study.

Exclusion Criteria:

Participants that meet any of the following criteria will be excluded from the trial:

1. Has a known or suspected allergy to components of the investigational product (e.g., cranberries, tart cherry, lemon balm, L-theanine).
2. Uncontrolled blood pressure or untreated hypertension.
3. Consumes >2 alcoholic beverages per day or >14 per week.
4. Major chronic illness or health condition that might interfere with the study outcomes at the discretion of the study clinician or principal investigator.
5. Use of antidepressant, anxiolytic, Central Nervous System stimulant, antipsychotic, antimanic, anti-inflammatory (except for aspirin and non-steroidal anti-inflammatory drugs [NSAIDS]. Multivitamins, vaccines, gender affirming hormones, HIV prevention medications, allergy medications, topical steroids are allowed for inclusion.)
6. Individuals who smoke or use nicotine patches or gum or e-cigarettes, or marijuana (within the past 6 months).
7. Individuals who have experienced a stroke or a head injury with concussion, loss of consciousness or seizures.
8. History or clinical manifestation of any significant neurologic disorder in the opinion of the investigator and/or study clinician.
9. Any disease, that by the investigator's judgement, could interfere with the intestinal barrier function, including Celiac disease (Lactose intolerance or acid reflux are allowed for inclusion).
10. Participants may not be receiving treatment involving experimental drugs. If the participant has been in a recent experimental trial, these must have been completed not less than one month prior to this trial.
11. Desire and/or plans on changing current diet and/or exercise regime during the participation of this trial.
12. Individuals who are pregnant or lactating.
13. Individuals currently of childbearing potential, but not using an effective method of contraception, as determined by the investigator.
14. History of heavy caffeinated beverage consumption (>400 mg caffeine/day - or 4 cups of coffee per day) within past 2 weeks prior to the Screening Visit (V1), or before their Baseline Visit (V2).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
To evaluate in healthy adults the effect of 7-day consumption of cranberry beverages compared to placebo on attention. | 7 days
  Change in Accuracy of Attention and Change in Speed of Attention composite scores outcomes from Baseline to each treatment phase (V3-8), assessed using the COMPASS cognitive assessment tool.

SECONDARY OUTCOMES:
To evaluate in healthy adults the effect of 7-day consumption of cranberry beverages compared to placebo on measures of focus. | 7 days
  Change in Overall % accuracy scores outcomes from Baseline to each treatment phase (V3-8), assessed using the STROOP task in the COMPASS cognitive assessment tool.
To evaluate in healthy adults the effect of 7-day consumption of cranberry beverages compared to placebo on measures of alertness. | 7 days
  Change in Alertness scores outcomes from Baseline to each treatment phase (V3-8), assessed using the self-rated Alertness Visual Analogue Scale in the COMPASS cognitive assessment tool.
To evaluate in healthy adults the effect of 7-day consumption of cranberry beverages compared to placebo on measures of cognition (accuracy of performance). | 7 days
  Change in Accuracy of Performance composite scores outcomes from Baseline to each treatment phase (V3-8), assessed using the COMPASS cognitive assessment tool.
To evaluate in healthy adults the effect of 7-day consumption of cranberry beverages compared to placebo on measures of cognition (speed of performance). | 7 days
  Change in Speed of Performance composite scores outcomes from Baseline to each treatment phase (V3-8), assessed using the COMPASS cognitive assessment tool.
To evaluate in healthy adults the effect of 7-day consumption of cranberry beverages compared to placebo on mood. | 7 days
  Change in Total Mood Disturbance scores from Baseline to each subsequent visit (V3-8), assessed using the Profile of Mood States-Short Questionnaire.
To evaluate in healthy adults the effect of 7-day consumption of cranberry beverages compared to placebo on stress. | 7 days
  Change in salivary cortisol from Baseline to each treatment phase (V3-8).

OTHER OUTCOMES:
To evaluate in healthy adults the safety and tolerability of 7-day consumption of cranberry beverages compared to placebo (Proportion of Adverse Events). | 7 days
  Proportion of Adverse Events per treatment phase by product causality.
To evaluate in healthy adults the safety and tolerability of 7-day consumption of cranberry beverages compared to placebo (Incidence of Adverse Events). | 7 days
  Incidence of mild, moderate, and severe Adverse Events per treatment phase by product causality.
To evaluate in healthy adults the safety and tolerability of 7-day consumption of cranberry beverages compared to placebo (Incidence of Serious Adverse Events). | 7 days
  Incidence of Serious Adverse Events per treatment phase by product causality.
To evaluate in healthy adults the safety and tolerability of 7-day consumption of cranberry beverages compared to placebo (Blood Pressure). | 7 days
  Change in Blood Pressure from Baseline to each subsequent visit (V3-8).
To evaluate in healthy adults the safety and tolerability of 7-day consumption of cranberry beverages compared to placebo (Heart Rate). | 7 days
  Change in Heart Rate from Baseline to each subsequent visit (V3-8).
To evaluate in healthy adults the safety and tolerability of 7-day consumption of cranberry beverages compared to placebo (Body Temperature). | 7 days
  Change in Body Temperature from Baseline to each subsequent visit (V3-8).

CONTACTS AND LOCATIONS:
Overall Officials: Alice Eggleston, PA-C, MPH, Principal Investigator — Atlantia Clinical Trials Ltd.
Locations (1):
- Atlantia Clinical Trials Ltd, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Travica N, D'Cunha NM, Naumovski N, Kent K, Mellor DD, Firth J, Georgousopoulou EN, Dean OM, Loughman A, Jacka F, Marx W. The effect of blueberry interventions on cognitive performance and mood: A systematic review of randomized controlled trials. Brain Behav Immun. 2020 Mar;85:96-105. doi: 10.1016/j.bbi.2019.04.001. Epub 2019 Apr 15. PMID 30999017
- [Result] Lamport DJ, Williams CM. Polyphenols and Cognition In Humans: An Overview of Current Evidence from Recent Systematic Reviews and Meta-Analyses. Brain Plast. 2021 Feb 9;6(2):139-153. doi: 10.3233/BPL-200111. PMID 33782647
- [Result] Scholey A, Gibbs A, Neale C, Perry N, Ossoukhova A, Bilog V, Kras M, Scholz C, Sass M, Buchwald-Werner S. Anti-stress effects of lemon balm-containing foods. Nutrients. 2014 Oct 30;6(11):4805-21. doi: 10.3390/nu6114805. PMID 25360512
- [Result] Kennedy DO, Scholey AB, Tildesley NT, Perry EK, Wesnes KA. Modulation of mood and cognitive performance following acute administration of Melissa officinalis (lemon balm). Pharmacol Biochem Behav. 2002 Jul;72(4):953-64. doi: 10.1016/s0091-3057(02)00777-3. PMID 12062586
- [Result] Kennedy DO, Little W, Scholey AB. Attenuation of laboratory-induced stress in humans after acute administration of Melissa officinalis (Lemon Balm). Psychosom Med. 2004 Jul-Aug;66(4):607-13. doi: 10.1097/01.psy.0000132877.72833.71. PMID 15272110
- [Result] Chai SC, Jerusik J, Davis K, Wright RS, Zhang Z. Effect of Montmorency tart cherry juice on cognitive performance in older adults: a randomized controlled trial. Food Funct. 2019 Jul 17;10(7):4423-4431. doi: 10.1039/c9fo00913b. PMID 31287117
- [Result] Yokogoshi H, Kobayashi M, Mochizuki M, Terashima T. Effect of theanine, r-glutamylethylamide, on brain monoamines and striatal dopamine release in conscious rats. Neurochem Res. 1998 May;23(5):667-73. doi: 10.1023/a:1022490806093. PMID 9566605
- [Result] Williams JL, Everett JM, D'Cunha NM, Sergi D, Georgousopoulou EN, Keegan RJ, McKune AJ, Mellor DD, Anstice N, Naumovski N. The Effects of Green Tea Amino Acid L-Theanine Consumption on the Ability to Manage Stress and Anxiety Levels: a Systematic Review. Plant Foods Hum Nutr. 2020 Mar;75(1):12-23. doi: 10.1007/s11130-019-00771-5. PMID 31758301